CLINICAL TRIAL: NCT04675151
Title: Safety and Efficacy of Nyxol (0.75% Phentolamine Ophthalmic Solution) With Pilocarpine Eye Drops in Subjects With Presbyopia
Brief Title: Safety and Efficacy of Nyxol With Pilocarpine Eye Drops in Subjects With Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPI-NYXP-201 (VEGA-1)
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2023-06

CONDITIONS: Presbyopia
Keywords: Nyxol; Presbyopia; Pilocarpine
MeSH Terms: conditions — Presbyopia | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nyxol + Pilocarpine (Experimental): 1 drop of Nyxol (Treatment 1) and 1 drop of Pilocarpine (Treatment 2)
  Interventions: Drug: Phentolamine Ophthalmic Solution 0.75%; Drug: Pilocarpine
- Nyxol (Active Comparator): 1 drop of Nyxol (Treatment 1)
  Interventions: Drug: Phentolamine Ophthalmic Solution 0.75%
- Pilocarpine (Active Comparator): 1 drop of Pilocarpine (Treatment 2)
  Interventions: Drug: Pilocarpine; Other: Placebo
- Placebo (Placebo Comparator): 1 drop of Placebo (Treatment 1)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phentolamine Ophthalmic Solution 0.75% — 0.75% phentolamine ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol; Nyxol®
  Arms: Nyxol; Nyxol + Pilocarpine
Drug: Pilocarpine — Pilocarpine ophthalmic solution
  Arms: Nyxol + Pilocarpine; Pilocarpine
Other: Placebo — Topical sterile ophthalmic solution
  Other Names: Phentolamine Ophthalmic Solution Vehicle
  Arms: Pilocarpine; Placebo

SUMMARY:
The objectives of this study are:

To evaluate the efficacy of Nyxol + Pilocarpine to improve DCNVA in subjects with presbyopia

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 40 and ≤ 64years of age.
2. BCDVA of 0.0 LogMAR(20/20 Snellen equivalent) or better in each eye under photopic conditions.
3. DCNVA of 0.4 LogMAR (20/50 Snellen equivalent) or worse under photopic conditions in each eye and binocularly.
4. Subjects who depend on reading glasses or bifocals in which their binocular best-corrected near VA is 0.1 LogMAR (20/25 Snellen equivalent) or better.

Exclusion Criteria:

Ophthalmic (in either eye):

1. Use of any topical prescription or OTC ophthalmic medications of any kind within 7 days of Screening until study completion.
2. Use of any over-the-counter (OTC) artificial tears (preserved or unpreserved) at least once per day within 7 days of Screening until study completion.
3. Current use of any topical ophthalmic therapy for dry eye.
4. Tear break-up time of < 5 seconds or corneal fluorescein staining.
5. Clinically significant ocular disease that might interfere with the study as deemed by the Investigator.
6. Recent or current evidence of ocular infection or inflammation in either eye.
7. Any history of herpes simplex or herpes zoster keratitis.
8. History of diabetic retinopathy or diabetic macular edema.
9. Known allergy, hypersensitivity, or contraindication to any component of the phentolamine, pilocarpine, or vehicle formulations.
10. History of cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal.
11. Ocular trauma, ocular surgery, ocular laser treatment within the 6 months prior to Screening. Any subject with multifocal intraocular lenses are excluded.
12. History of any traumatic (surgical or nonsurgical) or non traumatic condition affecting the pupil or iris.
13. Unwilling or unable to discontinue use of contact lenses.
14. Conjunctival hyperemia ≥ grade 2 on the CCLRU 4-point scale.

    Systemic:
15. Known hypersensitivity or contraindication to alpha- and/or beta adrenoceptor antagonists.
16. Known hypersensitivity or contraindication to any systemic cholinergic parasympathomimetic agents.
17. Clinically significant systemic disease that might interfere with the study as deemed by the Investigator.
18. Participation in any investigational study within 30 days prior to Screening.
19. Females of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.
20. Resting HR outside the specified range of 50 to 110 beats per minute.
21. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Clinical Site 12, Laguna Hills, California
  - Clinical Site 6, Newport Beach, California
  - Clinical Site 13, Crystal River, Florida
  - Clinical Site 5, Longwood, Florida
  - Clinical Site 11, Maitland, Florida
  - Clinical Site 8, Sarasota, Florida
  - Clinical Site 10, Roswell, Georgia
  - Clinical Site 3, Pittsburg, Kansas
  - Clinical Site 18, St Louis, Missouri
  - Clinical Site 16, Poughkeepsie, New York
  - Clinical Site 14, Fargo, North Dakota
  - Clinical Site 2, Athens, Ohio
  - Clinical Site 9, Cincinnati, Ohio
  - Clinical Site 7, Cleveland, Ohio
  - Clinical Site 15, Powell, Ohio
  - Clinical Site 4, Warwick, Rhode Island
  - Clinical Site 1, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- POS 0.75% First, Then LDP 0.4%: Participants received Phentolamine Ophthalmic Solution 0.75%: 0.75% phentolamine ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist, starting on the night of Visit 1 and subsequently taken daily for 3 to 4 consecutive days immediately prior to Visit 2.
  Then, after 3-4 days of initial administration of 0.75% POS, participants received Low-Dose Pilocarpine: 0.4% Pilocarpine ophthalmic solution, a direct-acting cholinergic agonist at Visit 2.
  Treatment 1 (0.75% POS) was administered in both eyes (OU) by the subject. Treatment 2 (0.4% LDP) was administered OU by a designated, unmasked site staff member, distinct from the site staff member recording assessments.
- POS 0.75% First, Then LDP Vehicle: Participants received Phentolamine Ophthalmic Solution 0.75%: 0.75% phentolamine ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist, starting on the night of Visit 1 and subsequently taken daily for 3 to 4 consecutive days immediately prior to Visit 2.
  Then, after 3-4 days of initial administration of 0.75% POS, participants received Low-Dose Pilocarpine Vehicle (Placebo): Topical Sterile Ophthalmic Solution at Visit 2.
  Treatment 1 (Nyxol or placebo) was administered in both eyes (OU)by the subject. Treatment 2 was administered OU by a designated, unmasked site staff member, distinct from the site staff member recording assessments.
  Treatment 1 (0.75% POS) was administered in both eyes (OU) by the subject. Treatment 2 (LDP Vehicle) was administered OU by a designated, unmasked site staff member, distinct from the site staff member recording assessments.
- POS Vehicle First, Then LDP 0.4%: Participants received Phentolamine Ophthalmic Solution Vehicle (Placebo): Topical Sterile Ophthalmic Solution, starting on the night of Visit 1 and subsequently taken daily for 3 to 4 consecutive days immediately prior to Visit 2.
  Then, after 3-4 days of initial administration of POS Vehicle, participants received Low-Dose Pilocarpine: 0.4% Pilocarpine ophthalmic solution, a direct-acting cholinergic agonist at Visit 2.
  Treatment 1 (Nyxol or placebo) was administered in both eyes (OU)by the subject. Treatment 2 was administered OU by a designated, unmasked site staff member, distinct from the site staff member recording assessments.
  Treatment 1 (POS Vehicle) was administered in both eyes (OU) by the subject. Treatment 2 (0.4% LDP) was administered OU by a designated, unmasked site staff member, distinct from the site staff member recording assessments.
- POS Vehicle First, Then LDP Vehicle: Participants received Phentolamine Ophthalmic Solution Vehicle (Placebo): Topical Sterile Ophthalmic Solution, starting on the night of Visit 1 and subsequently taken daily for 3 to 4 consecutive days immediately prior to Visit 2.
  Then, after 3-4 days of initial administration of POS Vehicle, participants received Low-Dose Pilocarpine Vehicle (Placebo): Topical Sterile Ophthalmic Solution at Visit 2.
  Treatment 1 (POS Vehicle) was administered in both eyes (OU) by the subject. Treatment 2 (LDP Vehicle) was administered OU by a designated, unmasked site staff member, distinct from the site staff member recording assessments.
Period: Overall Study
Arm/Group | POS 0.75% First, Then LDP 0.4% | POS 0.75% First, Then LDP Vehicle | POS Vehicle First, Then LDP 0.4% | POS Vehicle First, Then LDP Vehicle
Started | 44 | 30 | 31 | 45
Completed | 43 | 30 | 31 | 44
Not Completed | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | POS 0.75% First, Then LDP 0.4% | POS 0.75% First, Then LDP Vehicle | POS Vehicle First, Then LDP 0.4% | POS Vehicle First, Then LDP Vehicle | Total
Number analyzed (Participants) | 43 | 30 | 31 | 44 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (5.63) | 52.8 (5.11) | 52.7 (5.21) | 53.2 (4.55) | 53.1 (5.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 23 | 18 | 29 | 108
  Male | 5 | 7 | 13 | 15 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 4 | 10
  Not Hispanic or Latino | 42 | 27 | 29 | 40 | 138
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 3 | 3 | 1 | 4 | 11
  White | 40 | 26 | 28 | 38 | 132
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Study eye, n (%) [Count of Participants; unit: Participants]
  OD | 29 | 23 | 23 | 35 | 110
  OS | 14 | 7 | 8 | 9 | 38
Iris color, n (%) [Count of Participants; unit: Participants]
  Light blue | 5 | 6 | 3 | 6 | 20
  Dark blue | 0 | 2 | 2 | 3 | 7
  Blue with peripupillary brown | 14 | 5 | 7 | 9 | 35
  Uniform green | 1 | 1 | 3 | 4 | 9
  Green with brown iris ring | 5 | 4 | 4 | 4 | 17
  Central brown and peripheral green | 8 | 4 | 2 | 1 | 15
  Brown with some peripheral green | 3 | 2 | 5 | 4 | 14
  Brown | 7 | 6 | 5 | 13 | 31
Irides type, n (%) [Count of Participants; unit: Participants]
  Light | 25 | 18 | 19 | 26 | 88
  Dark | 18 | 12 | 12 | 18 | 60
Baseline photopic BCDVA study eye, letters read [Mean (Standard Deviation); unit: letters read at 4 m distance] | 57.8 (3.46) | 57.9 (2.84) | 58.1 (3.00) | 59.2 (3.58) | 58.3 (3.31)
Baseline photopic BCDVA fellow eye [Mean (Standard Deviation); unit: letters read at 4 m distance] | 58.5 (3.12) | 58.9 (3.39) | 57.7 (3.29) | 59.3 (3.69) | 58.7 (3.40)
Baseline photopic BCDVA binocular [Mean (Standard Deviation); unit: letters read at 4 m distance] | 61.0 (2.97) | 61.2 (3.53) | 60.0 (3.77) | 61.4 (3.560) | 60.9 (3.45)
Baseline mesopic BCDVA study eye [Mean (Standard Deviation); unit: letters read at 4 m distance] | 51.0 (3.95) | 49.5 (6.44) | 50.6 (5.83) | 52.2 (5.31) | 51.0 (5.36)
Baseline mesopic BCDVA fellow eye [Mean (Standard Deviation); unit: letters read at 4 m distance] | 51.3 (4.11) | 50.6 (6.53) | 50.2 (6.14) | 52.2 (5.06) | 51.2 (5.38)
Baseline mesopic BCDVA binocular [Mean (Standard Deviation); unit: letters read at 4 m distance] | 54.1 (3.31) | 54.2 (4.93) | 52.6 (5.44) | 54.8 (4.98) | 54.0 (4.68)
Baseline photopic DCNVA study eye [Mean (Standard Deviation); unit: letters read at 4 m distance] | 41.8 (5.39) | 37.9 (7.23) | 42.8 (5.34) | 42.0 (5.00) | 41.3 (5.90)
Baseline photopic DCNVA fellow eye [Mean (Standard Deviation); unit: letters read at 4 m distance] | 44.5 (4.48) | 42.8 (6.28) | 44.7 (4.61) | 44.9 (4.56) | 44.3 (4.95)
Baseline photopic DCNVA binocular [Mean (Standard Deviation); unit: letters read at 4 m distance] | 46.3 (3.85) | 45.3 (5.32) | 47.6 (3.49) | 46.1 (3.83) | 46.3 (4.15)
Baseline mesopic DCNVA study eye [Mean (Standard Deviation); unit: letters read at 4 m distance] | 36.2 (7.05) | 34.6 (6.81) | 37.3 (6.54) | 36.4 (6.45) | 36.2 (6.71)
Baseline mesopic DCNVA fellow eye [Mean (Standard Deviation); unit: letters read at 4 m distance] | 38.2 (6.59) | 37.3 (6.92) | 38.1 (6.35) | 37.3 (6.70) | 37.7 (6.59)
Baseline mesopic DCNVA binocular [Mean (Standard Deviation); unit: letters read at 4 m distance] | 41.4 (5.99) | 40.4 (6.36) | 40.1 (6.41) | 40.3 (6.05) | 40.6 (6.13)
Baseline photopic DCIVA study eye [Mean (Standard Deviation); unit: letters read] | 47.4 (6.87) | 45.3 (8.04) | 46.9 (6.34) | 46.0 (6.39) | 46.5 (6.86)
Baseline photopic DCIVA fellow eye [Mean (Standard Deviation); unit: letters read] | 48.7 (6.68) | 49.1 (7.01) | 48.4 (5.10) | 48.3 (6.19) | 48.6 (6.25)
Baseline photopic DCIVA binocular [Mean (Standard Deviation); unit: letters read] | 51.3 (6.42) | 52.6 (7.45) | 50.9 (4.87) | 51.5 (6.14) | 51.5 (6.24)
Baseline photopic PD study eye [Mean (Standard Deviation); unit: mm] | 4.297 (0.8347) | 4.494 (0.8190) | 4.342 (0.9966) | 4.265 (0.8782) | 4.337 (0.8756)
Baseline photopic PD fellow eye [Mean (Standard Deviation); unit: mm] | 4.267 (0.8277) | 4.608 (0.9048) | 4.391 (0.9617) | 4.340 (0.8299) | 4.384 (0.8731)
Baseline mesopic PD study eye [Mean (Standard Deviation); unit: mm] | 5.059 (0.8747) | 5.049 (0.7324) | 4.992 (1.1530) | 5.113 (0.8310) | 5.059 (0.8942)
Baseline mesopic PD fellow eye [Mean (Standard Deviation); unit: mm] | 5.136 (0.8759) | 5.100 (0.6839) | 4.996 (1.1266) | 5.197 (0.8201) | 5.117 (0.8789)
Baseline IOP study eye [Mean (Standard Deviation); unit: mmHg] | 14.4 (3.40) | 14.8 (3.14) | 13.9 (2.54) | 13.6 (2.88) | 14.1 (3.03)
Baseline IOP fellow eye [Mean (Standard Deviation); unit: mmHg] | 14.3 (2.99) | 14.9 (2.94) | 14.1 (2.41) | 13.8 (2.85) | 14.3 (2.83)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With ≥ 15 Letters of Improvement in Photopic Binocular DCNVA
Description: The primary efficacy endpoint was the percent of subjects with ≥ 15 letters of improvement in photopic binocular DCNVA on Visit 2 at 1 hour with POS + LDP compared to placebo alone. The improvement in binocular DCNVA for each subject was relative to the subject's own baseline value (Visit 1).
Time Frame: Visit 2 at 1 hour
Measure: Number; unit: percentage of subjects with ≥ 15 letters
Arm/Group | POS 0.75% First, Then LDP 0.4% | POS 0.75% First, Then LDP Vehicle | POS Vehicle First, Then LDP 0.4% | POS Vehicle First, Then LDP Vehicle
Number analyzed (Participants) | 43 | 30 | 31 | 44
percentage of subjects with ≥ 15 letters | 60.5 | 30.0 | 45.2 | 27.3

2. Secondary Outcome: Percentage of Subjects With Improvement of ≥ 5, ≥ 10, and ≥ 15 Letters in DCNVA (Photopic) From Baseline
Description: The percentage of subjects with improvement of ≥ 5, ≥ 10, and ≥ 15 letters in DCNVA (photopic) from Baseline at 0.5 hours, at 2 hours, at 3 hours, at 4 hours, and at 6 hours
Time Frame: Visit 2 at 0.5 hours, at 2 hours, at 3 hours, at 4 hours, and at 6 hours
Measure: Number; unit: percentage of subjects with improvement
Arm/Group | POS 0.75% First, Then LDP 0.4% | POS 0.75% First, Then LDP Vehicle | POS Vehicle First, Then LDP 0.4% | POS Vehicle First, Then LDP Vehicle
Number analyzed (Participants) | 43 | 30 | 31 | 44
percentage of subjects with improvement
  % of subjects with improvement of ≥ 5 letters from baseline at 0.5 hours | 88.4 | 86.7 | 74.2 | 70.5
  % of subjects with improvement of ≥ 10 letters from baseline at 0.5 hours | 76.7 | 50.0 | 54.8 | 52.3
  % of subjects with improvement of ≥ 15 letters from baseline at 0.5 hours | 60.5 | 33.3 | 25.8 | 15.9
  % of subjects with improvement of ≥ 5 letters from baseline at 2 hours | 88.4 | 93.3 | 83.9 | 70.5
  % of subjects with improvement of ≥ 10 letters from baseline at 2 hours | 81.4 | 60.0 | 71.0 | 45.5
  % of subjects with improvement of ≥ 15 letters from baseline at 2 hours | 62.8 | 26.7 | 41.9 | 18.2
  % of subjects with improvement of ≥ 5 letters from baseline at 3 hours | 95.3 | 83.3 | 83.9 | 72.7
  % of subjects with improvement of ≥ 10 letters from baseline at 3 hours | 67.4 | 60.0 | 64.5 | 43.2
  % of subjects with improvement of ≥ 15 letters from baseline at 3 hours | 46.5 | 26.7 | 48.4 | 20.5
  % of subjects with improvement of ≥ 5 letters from baseline at 4 hours | 95.3 | 83.3 | 83.9 | 75.0
  % of subjects with improvement of ≥ 10 letters from baseline at 4 hours | 67.4 | 60.0 | 51.6 | 50.0
  % of subjects with improvement of ≥ 15 letters from baseline at 4 hours | 46.5 | 30.0 | 32.3 | 20.5
  % of subjects with improvement of ≥ 5 letters from baseline at 6 hours | 88.4 | 86.7 | 71.0 | 72.7
  % of subjects with improvement of ≥ 10 letters from baseline at 6 hours | 67.4 | 60.0 | 54.8 | 50.0
  % of subjects with improvement of ≥ 15 letters from baseline at 6 hours | 37.2 | 36.7 | 22.6 | 18.2

3. Secondary Outcome: Percentage of Subjects With Improvement of ≥ 15 Letters in DCNVA (Photopic) at 1 Hour and With < 5 Letters of Loss in Photopic Binocular BCDVA From Baseline
Description: The percentage of subjects with improvement of ≥ 15 letters in DCNVA (photopic) at 1 hour and with < 5 letters of loss in photopic binocular BCDVA from Baseline
Time Frame: Visit 2 at 1 hour
Measure: Number; unit: % of subjects with improvement
Arm/Group | POS 0.75% First, Then LDP 0.4% | POS 0.75% First, Then LDP Vehicle | POS Vehicle First, Then LDP 0.4% | POS Vehicle First, Then LDP Vehicle
Number analyzed (Participants) | 43 | 30 | 31 | 44
% of subjects with improvement | 60.5 | 30.0 | 41.9 | 27.93

4. Secondary Outcome: Percentage of Subjects With Improvement in DCIVA (Photopic) From Baseline
Description: The percentage of subjects with improvement in DCIVA (photopic) from Baseline of ≥ 5, ≥ 10, and ≥ 15 letters
Time Frame: Visit 2 at 1 hour, at 3 hours, and at 6 hours
Measure: Number; unit: percentage with improvement
Arm/Group | POS 0.75% First, Then LDP 0.4% | POS 0.75% First, Then LDP Vehicle | POS Vehicle First, Then LDP 0.4% | POS Vehicle First, Then LDP Vehicle
Number analyzed (Participants) | 43 | 30 | 31 | 44
percentage with improvement
  % of subjects with improvement of ≥ 5 letters from baseline at 1 hour | 86.0 | 46.7 | 71.0 | 56.8
  % of subjects with improvement of ≥ 10 letters from baseline at 1 hour | 48.8 | 23.3 | 45.2 | 25.0
  % of subjects with improvement of ≥ 15 letters from baseline at 1 hour | 14.0 | 10.0 | 22.6 | 4.5
  % of subjects with improvement of ≥ 5 letters from baseline at 3 hours | 69.8 | 43.3 | 67.7 | 50.0
  % of subjects with improvement of ≥ 10 letters from baseline at 3 hours | 41.9 | 30.0 | 41.9 | 25.0
  % of subjects with improvement of ≥ 15 letters from baseline at 3 hours | 18.6 | 10.0 | 22.6 | 4.5
  % of subjects with improvement of ≥ 5 letters from baseline at 6 hours | 72.1 | 56.7 | 38.7 | 47.7
  % of subjects with improvement of ≥ 10 letters from baseline at 6 hours | 30.2 | 16.7 | 29.0 | 18.2
  % of subjects with improvement of ≥ 15 letters from baseline at 6 hours | 14.0 | 10.0 | 12.9 | 4.5

ADVERSE EVENTS:
Time Frame: 9 days.
Description: Data is not provided for each intervention separately as analyses by specific intervention were not conducted.
Arm/Group | POS 0.75% First, Then LDP 0.4% | POS 0.75% First, Then LDP Vehicle | POS Vehicle First, Then LDP 0.4% | POS Vehicle First, Then LDP Vehicle
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/30 | 0/31 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/30 | 0/31 | 0/45
Other Adverse Events (participants affected / at risk) | 15/44 | 6/30 | 6/31 | 2/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS 0.75% First, Then LDP 0.4% (N=44) | POS 0.75% First, Then LDP Vehicle (N=30) | POS Vehicle First, Then LDP 0.4% (N=31) | POS Vehicle First, Then LDP Vehicle (N=45)
Instillation site erythema (General disorders) | 6 (6) | 3 (3) | 2 (2) | 0 (0)
Installation site pain (General disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Installation site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Corneal dystrophy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT04675151/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04675151/SAP_001.pdf